CLINICAL TRIAL: NCT01905111
Title: An Open-label Phase I Dose Finding Study of BI 853520 Administered Orally in a Continuous Dosing Schedule in Japanese and Taiwanese Patients With Various Advanced or Metastatic Solid Tumours
Brief Title: A Study of BI 853520 in Japanese and Taiwanese Patients With Various Types of Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1300.15
Record Dates: First submitted 2013-07-12; First posted 2013-07-23 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (1):
- BI 853520 (Experimental): BI 853520 once daily in a dose escalation schedule
  Interventions: Drug: BI 853520

INTERVENTIONS:
Drug: BI 853520 — BI 853520 once daily in a dose escalation schedule

SUMMARY:
The primary objective of this trial is to explore the safety and tolerability of BI 853520 monotherapy and determine the maximum tolerated dose (MTD) for Japanese and Taiwanese patients with advanced or metastatic solid tumours.

Secondary objective is collection of preliminary data on anti-tumour efficacy

ELIGIBILITY:
Inclusion criteria:

* Patients with a confirmed diagnosis of advanced, measurable or evaluable, non-resectable and/or metastatic non-hematologic malignancy, which has shown to be progressive in the last 6 months
* Patients who have failed conventional treatment or for whom no therapy of proven efficacy exists or who are not amenable to established treatment options
* Recovery from reversible toxicities (alopecia excluded) of prior anti-cancer therapies (Common Terminology Criteria for Adverse Events grade <2)
* Age >= 20 years
* Written informed consent in accordance with International Conference on Harmonisation/Good Clinical Practice (ICH/GCP) and local legislation
* Eastern Cooperative Oncology Group (ECOG), performance score 0-1

Exclusion criteria:

* Serious concomitant non-oncological disease/illness
* Active/symptomatic brain metastases
* Second malignancy
* Pregnancy or breastfeeding
* Women or men who are sexually active and unwilling to use a medically acceptable method of contraception.
* Treatment with cytotoxic anti-cancer-therapies or investigational drugs within four weeks of the first treatment with the study medication

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Determination of the MTD. It will be defined by the occurrence of dose-limiting toxicities (DLT) during the first treatment cycle of each patient | After the first 28 days of treatment

SECONDARY OUTCOMES:
Objective response rate | Every 8 weeks until end of study participation, assessed up to 12 months
Disease control rate | Every 8 weeks until end of study participation, assessed up to 12 months
Duration of disease control | Every 8 weeks until end of study participation, assessed up to 12 months
Tumour shrinkage (in millimetre) defined as the difference between the minimum post-baseline sum of longest diameters of target lesions and the baseline sum of longest diameters of the same set of target lesions | Every 8 weeks until end of study participation, assessed up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- 1300.15.81001 Boehringer Ingelheim Investigational Site, Kashiwa-shi, Chiba, Japan
- 1300.15.88601 Boehringer Ingelheim Investigational Site, Taipei, Taiwan

REFERENCES:
- [Derived] Doi T, Yang JC, Shitara K, Naito Y, Cheng AL, Sarashina A, Pronk LC, Takeuchi Y, Lin CC. Phase I Study of the Focal Adhesion Kinase Inhibitor BI 853520 in Japanese and Taiwanese Patients with Advanced or Metastatic Solid Tumors. Target Oncol. 2019 Feb;14(1):57-65. doi: 10.1007/s11523-019-00620-0. PMID 30725402